CLINICAL TRIAL: NCT04750018
Title: Influence of Co-Vid 19 Pandemic on Screening Mammography in a Single Institution
Brief Title: Influence of Co-Vid 19 Pandemic on Screening Mammography Single Institution
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chen-Pin Chou (Other)
Responsible Party: Sponsor-Investigator, Chen-Pin Chou, Radiologist, Kaohsiung Veterans General Hospital.
Organization: Kaohsiung Veterans General Hospital. (Other)
Other Study IDs: KSVGH20-CT7-26
Record Dates: First submitted 2021-02-06; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: COVID-19; Breast Cancer
Keywords: COVID-19; Breast Cancer
MeSH Terms: conditions — COVID-19; Breast Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 2019: Patients receiving biopsies with a BI-RADS assessment of 4 or 5 from mammographic or ultrasonographic exams or combinations of tests were analyzed [4]. We further categorized the biopsy data as ultrasound-guided or mammograph-guided biopsy based on procedure coding. Ultrasound-guided core needle biopsy (CNB) was performed for breast lesions visible on ultrasound.
- COVID-19 2020: Patients receiving biopsies with a BI-RADS assessment of 4 or 5 from mammographic or ultrasonographic exams or combinations of tests were analyzed [4]. We further categorized the biopsy data as ultrasound-guided or mammograph-guided biopsy based on procedure coding. Ultrasound-guided core needle biopsy (CNB) was performed for breast lesions visible on ultrasound.
  Interventions: Other: surgery

INTERVENTIONS:
Other: surgery — Patients were divided into surgery and no disease.
  Groups: COVID-19 2020

SUMMARY:
To assess whether the COVID-19 pandemic delayed breast cancer diagnosis in Taiwan, an Asian country with a low COVID-19 incidence.

DETAILED DESCRIPTION:
The institutional review board approved this retrospective study at a public academic medical center. The monthly volume of breast biopsies and breast cancers during the COVID-19 pandemic (between January 1 and July 31, 2020) was compared to the same period a year earlier (pre-COVID-19).

ELIGIBILITY:
Inclusion Criteria:

* Receiving breast exam 2019-2020

Exclusion Criteria:

* lost clinical follow-up

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The test period of the COVID-19 pandemic was between January 1 and July 31, 2020. Moreover, the control period of the pre-COVID-19 pandemic was between January 1 and July 31, 2019, before there was any report about the virus. Only patients with complete medical records were eligible for enrollment in this study. Confirmed COVID-19 case numbers in Taiwan were acquired from Taiwan's National Health Command Center [7]. Anonymized records of breast biopsies and cancer registration in a single institution in southern Taiwan in the pre-COVID-19 and COVID-19 periods were reviewed.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-07-03 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
breast cancer | 1 year
  Breast cancer or not

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Pin Chou, MD, Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (1):
- Radiology depart, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on reasonable request from the corresponding author. Some data are not publicly available due to their containing information that could compromise the privacy of research participants.

REFERENCES:
- [Result] Chou CP, Pan HB, Yang TL, Chiang CL, Huang JS, Tsai MY. Impact of the COVID-19 pandemic on the volume of mammography examinations in Southern Taiwan. Breast J. 2021 Jan;27(1):89-91. doi: 10.1111/tbj.14019. Epub 2020 Aug 20. No abstract available. PMID 32815587
- [Derived] Chou CP, Lin HS. Delayed Breast Cancer Detection in an Asian Country (Taiwan) with Low COVID-19 Incidence. Cancer Manag Res. 2021 Jul 28;13:5899-5906. doi: 10.2147/CMAR.S314282. eCollection 2021. PMID 34349563